CLINICAL TRIAL: NCT04113824
Title: The Efficacy and Safety of Trapezius MSAT on Inpatients With Acute Whiplash Injury Caused by Traffic Accidents: A Randomized Controlled Trials
Brief Title: The Efficacy and Safety of Trapezius MSAT on Acute Whiplash Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JS-CT-2019-06
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Whiplash Injury of Cervical Spine; Neck Pain, Posterior
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: double blind, randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trapezius motion style acupuncture treatment (Experimental): The MSAT group recieved 3 sessions of MSAT; on second, third, fourth day after hospitalization. A trained doctor of Korean medicine with at least 3 years of clinical experience conducted the MSAT.
  The MSAT group were also treated with other Korean medical treatment everyday: acupuncture, chuna, pharmacoacupuncture and Korean herbal medicine.
  Interventions: Procedure: trapezuis motion style acupuncture treatment; Procedure: other Korean medical treatment
- Korean medical treatment (Active Comparator): The control group were received Korean medical treatment everyday after hospitalization: acupuncture, chuna, pharmacoacupuncture and Korean herbal medicine.
  Interventions: Procedure: other Korean medical treatment

INTERVENTIONS:
Procedure: trapezuis motion style acupuncture treatment — Motion Style Acupuncture Treatment(MSAT) is a therapeutic technique using acupuncture needle created in Jaseng Hospital. This treatment involves patients with musculoskeletal pain to move the part of their body actively during acupuncture treatment under physicians' observation
  Arms: trapezius motion style acupuncture treatment
Procedure: other Korean medical treatment — acupuncture treatment, chuna, pharmacoacupuncture, Korean herbal medicine

SUMMARY:
This study is a double blind, randomized controlled trail. condition/disease: acute neck pain treatment/intervention: motion style acupuncture treatment

DETAILED DESCRIPTION:
Motion Style Acupuncture Treatment(MSAT) is a therapeutic technique using acupuncture needle created in Jaseng Hospital. This treatment involves patients with musculoskeletal pain to move the part of their body actively during acupuncture treatment under physicians' observation. This treatment is known to relieve the pain and increase the range of motion(ROM). However, there has been no specific value for the effect of this treatment.

So, we conducted a randomized controlled trials to verify the efficacy and safety of trapezuis MSAT. From July 2019 to September 2019, we collected 100 inpatients who were suffered from posterior nick pain with the numeric rating scale(NRS) over 4 after whiplash injury by acute traffic accident(TA). For experimental group(n=50), we conducted MSAT three times(on 2nd, 3rd and 4th day of hospitalization) and other Korean medical treatment. For control group(n=50), just Korean medical treatment except MSAT was conducted. For these two groups, we compared NRS, Visual Analogue Scale(VAS), Range Of Motion(ROM), Nthe amount of pain via NRS(Numeric Rating Scale), VAS(Visual Analogue Scale), ROM(Range Of Motion), Neck Disability Index (NDI), and EuroQol 5-Dimension (EQ-5D).

ELIGIBILITY:
Inclusion Criteria:

* Patients who needs hospitalization due to acute whiplash injury that occurred within 7 days after traffic accident
* Patients with NRS ≥ 5 for posterior neck pain
* Patients aged 19-70 years on the date they sign the consent form
* Patients who provide consent to participate in the trial and return the informed consent form

Exclusion Criteria:

* Patients with a specific serious disease that may cause spinal pain: malignancy, spondylitis, inflammatory spondylitis, etc.
* Patients with progressive neurological deficits or with severe neurological symptoms
* Patients who have had surgery or procedures within the last three weeks
* The cause of pain is due to soft tissue disease, not the spine: tumors, fibromyalgia, rheumatoid arthritis, gout, etc.
* Patients with other chronic conditions that may interfere with the interpretation of the therapeutic effects or results: cardiovascular disease, kidney disease, diabetic neuropathy, dementia, epilepsy, etc.
* Patients who are taking steroids, immunosuppressants, mental illness drugs, or other drugs that may affect the results of the study
* If acupuncture is inadequate or unsafe: patients with hemorrhagic, receiving anticoagulants, severe diabetes and cardiovascular disease
* Patients who are pregnant or planning to become pregnant
* Patients with a serious mental illness
* Patients who are participated in clinical trials other than observational studies without therapeutic intervention.
* Patients who are difficult to complete the research participation agreement
* Other patients whose participation in the trial is judged by a researcher to be problematic

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2019-09-07 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale(NRS) of neck pain | day 5
  The extent of posterior neck pain and discomfort was assessed using NRS. NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10. The participant is asked to report their posterior neck pain and discomfort using NRS, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) of neck pain | day 5
  VAS is an assessment index in which the patient records their pain on a 100mm line from 'no pain' at one end, and 'the most severe pain imaginable' at the other end.
Visual Analogue Scale (VAS) of arm pain | day 5
  VAS is an assessment index in which the patient records their pain on a 100mm line from 'no pain' at one end, and 'the most severe pain imaginable' at the other end.
Numeric Rating Scale(NRS) of arm pain | day 5
  NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10.
Physical examination (Cervical range of motion) | day 5
  ROM of flexion, extension, lateral flexion, rotation was measured.
Neck Disability Index (NDI) | day 5
  The Neck Disability Index (NDI) is a 10-item questionnaire that measures a patient's self-reported neck pain related disability.
EuroQol 5-Dimension (EQ-5D) | day 5
  The EQ-5D is a method of indirectly calculating the weights of certain health states for quality of life after a multidimensional investigation of health states, and is the most widely used instrument for this purpose. The EQ-5D consists of 5 questions about current health state (mobility, self-care, usual activities, pain, anxiety/depression), and each question is scored on a 5-point Likert scale (1=no problems, 3=moderate problems, 5=severe problems). In this study, we will use the Korean version of the EQ-5D, which has been demonstrated to be valid.
Patient Global Impression of Change (PGIC) | day 5
  The PGIC is an index that assesses improvements in functional limitation caused by whiplash injury. Participants rate the improvement in functional limitations after treatment on a 7-point Likert scale (1=Very much improved, 4=No change, 7=Very much worse). This index was originally developed for use in Psychology, but is currently used in various other medical fields to assess improvements in pain.
Drug Consumption | day 5
  Check drug consumption change every visit
Adverse events | day 5
  Check adverse events every visit

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, PhD, Study Chair — Jaseng Medical Foundation
Locations (2):
- South Korea (2):
  - Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu
  - Jaseng Medical Foundation, Seoul

IPD SHARING:
Plan to Share IPD: No